CLINICAL TRIAL: NCT05639803
Title: A Phase I，Randomized, Double-blind，Placebo Controlled，Dose Escalated, Single Adminstrated Clinical Trial of PEGIFNα1b in Chinese Healthy Adults
Brief Title: A Clinical Trial of PEGIFNα1b in Chinese Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SH-002-01
Record Dates: First submitted 2020-06-16; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Herpes Zoster
Keywords: Peginterferon α1b for Injection
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- PEGIFNα1b 1.5 μg/kg (Experimental): 8 randomized participants receive one dose PEGIFNα1b 1.5 μg/kg, 2 randomized participants receive one dose placebo, subcutaneous administered
  Interventions: Drug: PEGIFNα1b; Drug: Placebo
- PEGIFNα1b 3.0 μg/kg (Experimental): 8 randomized participants receive one dose PEGIFNα1b 3.0 μg/kg, 2 randomized participants receive one dose placebo, subcutaneous administered
  Interventions: Drug: PEGIFNα1b; Drug: Placebo
- PEGIFNα1b 5.0μg/kg (Experimental): 8 randomized participants receive one dose PEGIFNα1b 5.0 μg/kg, 2 randomized participants receive one dose placebo, subcutaneous administered
  Interventions: Drug: PEGIFNα1b; Drug: Placebo
- PEGIFNα1b 6.0 μg/kg (Experimental): 8 randomized participants receive one dose PEGIFNα1b 6.0 μg/kg, 2 randomized participants receive one dose placebo, subcutaneous administered
  Interventions: Drug: PEGIFNα1b; Drug: Placebo
- PEGIFNα1b 7.0 μg/kg (Experimental): 8 randomized participants receive one dose PEGIFNα1b 7.0 μg/kg, 2 randomized participants receive one dose placebo, subcutaneous administered
  Interventions: Drug: PEGIFNα1b; Drug: Placebo

INTERVENTIONS:
Drug: PEGIFNα1b — 100μg/vial
Drug: Placebo — 0.5ml/vial

SUMMARY:
This is a Phase I，randomized, double-blind, placebo controlled,dose escalated,single administrated clinical trial in Chinese healthy adult's volunteers.

In the trial, it is planned to enroll 50 subjects, randomized to 5 dosage groups to receive the test drug and the placebo control.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, dose-escalation, single-dose phase I clinical study, including safety tolerability assessment, pharmacokinetic studies and immunogenicity studies, to evaluate the expression level of mRNA in whole blood of 2',5'-oligoadenylate synthetase, as well as the level of Neopterin (NTP) in serum.

ELIGIBILITY:
Inclusion Criteria:

* Must agree to and voluntarily sign a written Informed Consent prior to the study.
* Must be healthy males or females.
* Between 18 to 70 years old, inclusive.
* Must have a body mass index (BMI) of 19 to 26 kg/m2, inclusive, and male subject must have a minimum body weight of 50.0 kg,female subject must have a minimum body weight of 45kg.

Exclusion Criteria:

* History of allergic or anaphylactic reactions or known allergy to any component of interferon medication including the study drug.
* Having abnormality in physical examination,vital signs, electrocardiogram,eye,skin(e.g., psoriasis,sarcoidosis) within screening and the abnormality is considered clinically significant as determined by the investigator.
* Laboratory values (platelet, hemoglobin or neutrophils)that were outside the normal range，ALT，AST or TG>1.5 fold normal range，positive test result for pregnancy,hepatitis B surface antigen(HBsAg) ,hepatitis C antibody (HCV Ab),treponema pallidum antibody or human immunodeficiency virus antibody(HIV Ab), thyroid function abnormal within screening.
* Having any ischemic disease,autoimmune disease,infectious disorders,history of neuropsychiatric disease (e.g., epilepsy,depression,suicidal behavior).
* History of any disease (gastrointestinal tract,renal,hepatic,neurologic,hematologic,endocrinologic, tumor, pulmonary, cardiovascular and/or other major disease), or organ transplantation within 6 months prior to screening.
* Unlikely to comply with unified diet or having difficulty to swallow.
* Treatment with any medication( prescription/nonpreserip drugs/vitamins/herbs ) within 30 days prior to screening.
* History of alcohol abuse (more than 14 units of alcohol per week, one unit of alcohol equals 360ml beer or 150ml wine or 45ml strong drinks containing 40% alcohol) within 3 months prior to screening or a positive screen test for presence for alcohol at screening or into hospital.
* Consuming any special diet(including dragon fruit,mango,grapefruit,etc. ) or doing strenuous exercise within 2 weeks prior to screening. Consuming alcohol or caffeine containing products(e.g., coffee,tea, coco,chocolate ) within 48 hours of dosing. Intaking any products can affecting drug absorption,distribution,excretion,metabolism.
* Regular smoking with consumption ≥ 5 cigarettes per day winthin 3 months prior to screening.
* Treatment with any interferon product within 6 months prior to screening.
* Participation in any other medication or device study within 3 months prior to screening.
* History of drug (morphine,marihuana,methamphetamine,dimethylamphetamine,ketamine,etc.) abuse or a positive screen test for presence for drugs.
* Having donated or lost 200 mL or more of blood within 3 months prior to screening or plan to donate blood throughout the study and within 3 months after the study.
* Lactating mothers,male subjects(or pairs) and female subjects have child-bearing/sperm or egg donation plan from 30 days before study to 3 months after study while unwill to practice effective birth control throughout the study.
* History of blood or needle phobia.
* Driving or operating delicated machinery throughout the study.
* Investigator discretion as to unsuitability

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2020-10-22 (Actual); Study Completion 2020-10-22 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | receive PEGIFNα1b (day 1) to day 28
  The number of adverse events associated with the PEGIFNα1b/placebo will be collected and measured.
λz | Receive PEGIFNα1b/placebo (day 1) to day 15.
  Pharmacokinetic assessments
Tmax | Receive PEGIFNα1b/placebo (day 1) to day 15.
  Pharmacokinetic assessments
Peak Plasma Concentration (Cmax) | Receive PEGIFNα1b/placebo (day 1) to day 15.
  Pharmacokinetic assessments
Area under the plasma concentration versus time curve (AUC) | Receive PEGIFNα1b/placebo (day 1) to day 15
  Pharmacokinetic assessments
ADA | Receive PEGIFNα1b/placebo (day 1) to day21.
  ADA in plasma of participants for immunogenicity assessments.
Nab | Receive PEGIFNα1b/placebo (day 1) to day21.
  Nab in plasma of participants for immunogenicity assessments.

SECONDARY OUTCOMES:
Level of Neopterin | Receive PEGIFNα1b/placebo (day 1) to day15
  Plasma concentration of 2',5'-OAS(Type I,II), Neopterin

CONTACTS AND LOCATIONS:
Overall Officials: Shanghai Institute Of Biological Products Co., Ltd, Study Director — SINOPHARM; The first affiliated hospital of bengbu medical college, Principal Investigator — Bengbu medical college
Locations (1):
- The first affiliated hospital of bengbu medical college, Bengbu, Anhui, China